CLINICAL TRIAL: NCT01928407
Title: A Phase IV, Prospective, Multicenter , Randomized Open Label, 48 Weeks Study to Evaluate the Antiretroviral Efficacy and Safety of Atazanavir or Darunavir,Each in Combination With a Fixed Dose of Tenofovir Emtricitabine in HIV-1-infected Treatment-naïve Subjects With CD4counts Below 200 µL.
Brief Title: Evaluation of the Efficacy and Safety Between Two Antiretroviral Regimens, in HIV-1-infected Treatment-naïve Subjects With Low CD4 Counts
Acronym: DATA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMEA 040-DATA
Record Dates: First submitted 2013-06-19; First posted 2013-08-26 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: HIV-1 Infection; Immunosuppression-related Infectious Disease
Keywords: naives, CD4 < 200 cell/mm3, Atazanavir, Darunavir
MeSH Terms: interventions — Darunavir; Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATAZANAVIR (Experimental): The patient included in this Group 1 will receive their first antiretroviral regimen included : ATV + TDF/FTC (or Abacavir/Lamivudine, [ABC/3TC], if contre indicated of TDF/FTC) The dose : atazanavir/ritonavir 300/100mg/day and TDF/FTC 245 /200 mg day, 3 pills once a day, during 48 weeks during a meal
  Interventions: Drug: ATAZANAVIR
- DARUNAVIR (Experimental): The patients included in this Group 2 will receive their first antiretroviral regimen included Group 2 : DRV+ TDF/FTC (or ABC/3TC if contre-indicated of TDF/FTC) The dose : darunavir/ritonavir 800/100mg/day and TDF/FTC 245 /200 mg day, 4 pills once a day, during 48 weeks during a meal
  Interventions: Drug: DARUNAVIR

INTERVENTIONS:
Drug: DARUNAVIR — The patient included will receive their first antiretroviral regimen included the darunavir treatment in combination with 2 others molecules
  Other Names: Prezista
  Arms: DARUNAVIR
Drug: ATAZANAVIR — The patient included will receive their first antiretroviral regimen included the atazanavir treatment in combination with 2 others molecules
  Other Names: REYATAZ
  Arms: ATAZANAVIR

SUMMARY:
A phase IV, prospective, multicenter , randomized open label, 48 weeks study to evaluate the antiretroviral efficacy and safety of atazanavir/ritonavir or darunavir/ritonavir, each in combination with a fixed dose of tenofovir disoproxil fumarate- emtricitabine in HIV-1-infected treatment-naïve subjects with CD4 counts below 200 µL.

DETAILED DESCRIPTION:
Principal objective

To evaluate the virological efficacy and safety at week 48 of 2 regimens atazanavir/ritonavir (ATZ/r) 300/100 mg or darunavir/ritonavir (DRV/r) 800/100 mg, each in combination with a fixed-dose of tenofovir/emtracitabine in HIV-1 treatment-naïve subjects with CD4 counts below 200 µL.

Secondary objectives

* Proportion of subjets with virologic efficacy at week 24
* Proportion of subjects with confirmed virologic failure at week 24 or later
* Proportion of patients with virologic mutations
* Evaluate the virologic effect in seminal fluid
* To evaluate immunological response over time up to week 48
* To assess plasma and seminal pharmacokinetics of the drugs in the treatment regimen at week 4, 24, and 48
* Correlate the pharmacokinetic properties of the drugs with virologic outcome in plasma and semen at week 4 and 48
* Correlate the free fraction (not bound to protein) of atazanavir and darunavir in plasma and semen to virologic outcome
* Evaluate the relationship of bilirubinemia with atazanavir
* Change from baseline in fasting lipids, fasting glucose and insulin over time in the 2 arms
* Compare adherence patient satisfaction and sexual behaviour between the regimens

Methodology

This is a 48 week, multicentre, prospective, open label, phase IV, randomized. non comparative, study.

Inclusion criteria

* Male or female, aged > 18 years of age.
* HIV-1 infection determined by a positive ELISA and confirmed by Western blot
* Plasma HIV-RNA > 1 000 c/mL
* CD4+T cell count < =200 cells/mm3 at the time of screening, or < =250 cells/mm3 if the CD4 count was <200 cells/mm3 12 weeks before screening.
* Women of childbearing potential must agree to use an effective method of barrier contraception or have documented sterility.
* Subjects must have medical insurance throught the Securite Sociale
* Ability to understand and provide written informed consent.

Non-inclusion criteria

* Acute opportunistic infection within the past two weeks
* HIV-2 infection
* pregnant woman
* Any subject with drug resistance mutations at screening
* Any subject with a grade 3 or greater clinical or laboratory adverse event at screening
* Any subject who has received antiretoviral therapy except for prevention of mother to child transmission and patients who has received post exposure prophylaxis for a a month or less
* calculated creatinine clearance < 60/mL as estimated by the Cockcroft- Gault equation
* Patients in the opinion of the investigator that are unlikley to be able to follow study instructions
* Any subject unable to take antiretroviral medication for whatever reason
* Any subject taking a treatment or medication that is contraindicated when co-administered with any arm or drug in the treatment.

Treatment:

* Group 1 : ATV + TDF/FTC (or Abacavir/Lamivudine, [ABC/3TC], if TDF/FTc contre-indicated
* atazanavir/ritonavir 300/100mg/day and TDF/FTC 245 /200 mg by day, 3 pills once a day, during 48 weeks during a meal
* Group 2 : DRV+ TDF/FTC (or ABC/3TC if TDF/FTc contre-indicated)
* darunavir/ritonavir 800/100mg/day and TDF/FTC 245 /200 mg by day, 4 pills once a day, during 48 weeks during a meal

Primary Endpoints :

* Proportion of patients with HIV-1 plasma viral load below 50 copies/mL at week 48 while receiving their initial regimen
* Proportion of patients experiencing grade 2-4 adverse clinical and laboratory events including hematology, chemistry, lipids (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides), glucose and insulin by week 48.

Secondary endpoints:

* Proportion of patients with plasma HIV RNA below 50 cp/mL at week 24
* Proportion of patients with HIV RNA> 50 cp/mL at week 24 or later confirmed by a second HIV RNA at least 14 days after the first test
* Development of resistance mutations in subjects who have virologic failure testing at 24 weeks or later tested by a genotypic resistance test
* Evaluate the virologic effect in seminal fluid at baseline, W4 and W48 by change in HIV RNA concentrations in semen over time
* To evaluate immunological response over time up to week 48 in the 2 arms by CD4 cell count ( W-4, W2,W4, W12, W36 and W48), differenciation and activation in T CD4 ( W2,W4, W12, W24 and W48); Change in lymphocyte subset reconsistution at week 48 compared to baseline. ; Change in immunolgic markers of inflammations at weeks 2, 4, 12, 24, 48
* To assess plasma and seminal pharmacokinetics of the drugs in the treatment regimen at week 4, 24, and 48 through residual concentrations ( C min) of antiretroviral drugs at W4, W24, and W48
* Atazanavir and darunavir (plasma and seminal) drug concentrations and coorelation with adverse clinical and laboratory events.
* Evaluate the relationship of bilirubinemia with atazanavir pharmacokinetics (Cmin)
* Evolution of lipid, glucose and insulin parameters from baseline to weeks 24 and 48
* Adherence to regimen, patient satisfaction and sexual behaviour between the regimens at W2,W24 and W48 mesured by ( mettre ref)
* Evolution of anthropomorphic measurements from baseline to weeks 24, 48.

Substudies Brief description (2 lines maximum) and person in charge of the substudy

* Immunologic substudy ( Pr Brigitte Autran) : Change in immunolgic markers of inflammations at weeks 2, 4, 12, 24, 48 and change in lymphocyte subset reconsistution at week 48 compared to baseline.
* Pharmacologic substudy ( Dr Gilles Peytavin) : To assess plasma and seminal pharmacokinetics of the drugs in the treatment regimen at week 4, 24, and 48 through residual concentrations ( C min) of antiretroviral drugs at W4, W24, and W48
* Virologic substudy ( Dr Anne Geneviève Marcelin) : Evaluate the virologic effect in seminal fluid at baseline, W4 and W48
* Behaviour substudy ( Dr France Lert) : Compare adherence patient satisfaction and sexual behaviour between the regimens at W2,W24 and W48

Estimated enrolment: 120 subjects (60 per group) randomly assigned 1:1

ELIGIBILITY:
Inclusion Criteria

* Male or female, aged > 18 years of age
* HIV-1 infection determined by a positive ELISA and confirmed by Western blot
* Plasma HIV-RNA > 1 000 c/mL
* CD4+T cell count < =200 cells/mm3 at the time of screening, or < =250 cells/mm3 if the CD4 count was <200 cells/mm3 12 weeks before screening
* Women of childbearing potential must agree to use an effective method of barrier contraception or have documented sterility
* Subjects must have medical insurance throught the Securite Sociale
* Ability to understand and provide written informed consent

Exclusion Criteria

* Acute opportunistic infection within the past two weeks
* HIV-2 infection
* Pregnant woman
* Any subject with drug resistance mutations at screening
* Any subject with a grade 3 or greater clinical or laboratory adverse event at screening
* Any subject who has received antiretoviral therapy except for prevention of mother to child transmission and patients who has received post exposure prophylaxis for a a month or less
* Calculated creatinine clearance < 60/mL as estimated by the Cockcroft- Gault equation
* Patients in the opinion of the investigator that are unlikley to be able to follow study instructions
* Any subject unable to take antiretroviral medication for whatever reason
* Any subject taking a treatment or medication that is contraindicated when co-administered with any arm or drug in the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02-23 (Actual); Primary Completion 2011-03-29 (Actual); Study Completion 2013-01-07 (Actual)

PRIMARY OUTCOMES:
Viral load of HIV-1 < 50 cp/ml | 48 weeks
  To evaluate the virological efficacy and safety at week 48 of 2 regimens atazanavir/ritonavir (ATZ/r) 300/100 mg or darunavir/ritonavir (DRV/r) 800/100 mg, each in combination with a fixed-dose of tenofovir/emtracitabine in HIV-1 treatment-naïve subjects with CD4 counts below 200 µL

SECONDARY OUTCOMES:
• Proportion of subjets with virologic efficacy | 24 weeks
  • Proportion of subjets with virologic efficacy (viral load of HIV-1 <50 cp/ml)
• Proportion of subjects with confirmed virologic failure | 24 weeks
  • Proportion of subjects with confirmed virologic failure (viral load > 50 cp/ml on 2 consecutive mesures)
Viral lod of HIV-1 on seminal fluid | W00,W4 et W48
  • Evaluate the viral load of HIV-1 at week 0, week 4 and week 48 on the seminal fluid (substudy)
Immunologic response | W-4,W2,W4,W12,W24 and W48
  • Evaluate the immunologic response by the CD4 mesearement at W-4,W2,W4,W12,W24 and W48
Differenciation and activation of lymphocytes | W0,W2,W4,W12,W24 and W48
  At the end of the study, in a central lab, we will measure some inflammation and activation markers (CD69, HLA-DR, CD38, annexine V, IL-6, CD14s, IL-7 plasma) of lymphocytes CD4 and CD8(with the plasmatheque collected during the study)
Pharmacokinetics evaluation of the drugs in plasma | W4,W24 and W48
  Measure of drugs (atazanir and darunavir) concentration (24 hours after taking treatment)in plasma at week 4, 24, and 48
Pharmacokinetic evaluation of the drugs in semen | W4 and W48
  Measure of drugs (atazanir and darunavir) concentration (24 hours after taking treatment)in semen at week 4 and 48
• Evaluate the relationship of bilirubinemia with atazanavir | W4 and W48
  Evaluate the relationship of the evolution of the measure of bilirubinemia (collected during study) with the concentration of atazanavir in blood
Fasting glucose, lipids and insulin | W48
  • Change from baseline in fasting lipids, fasting glucose and insulin over time in the 2 arms
Clinic and biologic tolerance | W48
  Evaluate the clinic and biologic tolerance between the 2 regimens (adverse event and some biologic measure will be collected for this evaluation).
  We will see in two arms if there are more adverse event or biological event.
Sexual behaviour | W0,W24 et W48
  • Compare sexual behaviour between the regimens (substudy with a questionnary)
Adherence patient satisfaction | W2,W24 et W48
  • Compare adherence patient satisfaction between the regimens (with questionnary)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence LS SLAMA, PhD, Principal Investigator — Hospital TENON; Roland RL LANDMAN, PhD, Principal Investigator — Institut de Médecine et d'Epidémiologie Appliquée - Fondation Internationale Léon M'Ba
Locations (29):
- France (29):
  - Hopital Zobda Quitman, Fort de France, Martinique
  - Centre Hospitalier D'Argenteuil, Argenteuil
  - Hopital Saint-Jacques, Besançon
  - Hopital Avicenne, Bobigny
  - Hopital Jean Verdier, Bondy
  - Hopital Saint-Andre, Bordeaux
  - Chu Cote de Nacre, Caen
  - Hopital Louis Mourier, Colombes
  - Hopital Le Bocage, Dijon
  - Hopital Raymond Poincare, Garches
  - C.H.D de Vendee, La Roche-sur-Yon
  - Hopital Dupuytren, Limoges
  - Hopital Sainte-Marguerite, Marseille
  - Centre Hospitalier de Melun, Melun
  - Hopital L'Archet, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Necker, Paris
  - Hopital Bichat, Paris
  - Hopital Tenon, Paris
  - Hopital Cochin, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint-Jean Roussillon, Perpignan
  - Hopital Rene Dubos, Pontoise
  - C.H.R.A, Pringy
  - Hopital Civil, Strasbourg
  - Hopital Gustave Dron, Tourcoing
  - Hopital Bretonneau, Tours

REFERENCES:
- [Derived] Slama L, Landman R, Assoumou L, Benalycherif A, Samri A, Joly V, Pialoux G, Valin N, Cabie A, Duvivier C, Lambert-Niclot S, Marcelin AG, Peytavin G, Costagliola D, Girard PM; IMEA 040 DATA Study Group. Efficacy and safety of once-daily ritonavir-boosted atazanavir or darunavir in combination with a dual nucleos(t)ide analogue backbone in HIV-1-infected combined ART (cART)-naive patients with severe immunosuppression: a 48 week, non-comparative, randomized, multicentre trial (IMEA 040 DATA trial). J Antimicrob Chemother. 2016 Aug;71(8):2252-61. doi: 10.1093/jac/dkw103. Epub 2016 Apr 10. PMID 27068399